CLINICAL TRIAL: NCT00905138
Title: Double Blind, Placebo-controlled Trial for the Assessment of Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Single Ascending and Multiple Oral Doses of GLPG0259 in Healthy Subjects
Brief Title: First-in-Human Single Ascending and Multiple Dose of GLPG0259
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos NV
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0259-CL-101
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): single ascending doses
  Interventions: Drug: GLPG0259
- 2 (Placebo Comparator): single dose placebo
  Interventions: Drug: placebo
- 3 (Experimental): multiple dose, 5 days, oral solution
  Interventions: Drug: GLPG0259
- 4 (Placebo Comparator): multiple dose, 5 days, oral solution
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GLPG0259 — single ascending doses, oral solution
  Arms: 1
Drug: placebo — single dose, oral solution
  Arms: 2
Drug: GLPG0259 — multiple dose, oral solution, 5 days
  Arms: 3
Drug: placebo — oral solution, 5 days
  Arms: 4

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) and multiple (MD) oral dose of GLPG0259 compared to placebo.

Also, pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0259 after single and multiple oral administration will be evaluated, and, if applicable, the maximum tolerated dose determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple dosing | up to 10 days postdose

SECONDARY OUTCOMES:
Pharmacokinetics of single and repeated doses | up to 10 days postdose
Exploratory evaluation of TNF-alpha and IL6 in whole blood | up to 12 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Johan Beetens, PharmD, PhD, Study Director — Galapagos NV; Eva Vets, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium